CLINICAL TRIAL: NCT00751426
Title: Treatment of Chronic Hepatitis c With Interferon-Alpha 2a and Ribavirin: a Comparison of Patients With Psychiatric Disorders and Controls
Brief Title: Treatment of Hepatitis C in Psychiatric Patients
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Martin Schaefer, MD
Other Study IDs: Psy 225/98
Record Dates: First submitted 2008-09-11; First posted 2008-09-12 (Estimated); Last update posted 2008-09-12 (Estimated); Status verified 2008-08

CONDITIONS: Mental Disorders; Drug Addiction
Keywords: Interferon-alpha; hepatitis c; Drug addiction; methadone; psychiatric disorder; Safety and efficacy of Interferon-alpha i patients with a psychiatric disorder.
MeSH Terms: conditions — Mental Disorders; Substance-Related Disorders; Hepatitis C

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Psychiatric disorders or drug addiction are often regarded as contraindications against the use of Interferon-alpha in patients with chronic hepatitis C. The investigators aim is/was to get prospective data about adherence, efficacy and mental side effects of IFN-alpha treatment in different psychiatric risk groups compared to controls. In a prospective trial, 81 patients with chronic hepatitis C (positive HCV-RNA and elevated ALT) and psychiatric disorders (n=16), methadone substitution (n=21), former drug addiction (n=21) or controls without psychiatric history or addiction (n=23) should be/were treated with a combination of IFN-alpha-2a 3 x 3 Mio U/week and ribavirin (1000-1200 mg/day).

DETAILED DESCRIPTION:
Patients from the Munich University outpatient department of psychiatry or gastroenterology as well as inpatients with elevated transaminases were tested for HCV-infection and considered for our trial to avoid a positive or negative selection. Medical inclusion criteria were a detectable serum HCV-RNA level in a PCR-based assay (AMPLICOR®, Roche Diagnostics, Branchburg, NJ) for more than 6 months and an elevated alanine aminotransferase (ALT > 30 U/L, normal <24 U/L). General exclusion criteria were the presence of other liver disease, Child B or C cirrhosis, severe cardiac or neurological disease, co-infection with hepatitis B or HIV, hepatocellular carcinoma evaluated by ultrasound and alpha-fetoprotein, autoimmune disorders, a neutrophil count below 1500 per cubic millimetre, and a platelet count below 75000 per cubic millimetre.

ELIGIBILITY:
Inclusion Criteria:

* Medical inclusion criteria were a detectable serum HCV-RNA level in a PCR-based assay (AMPLICOR®, Roche Diagnostics, Branchburg, NJ) for more than 6 months and an elevated alanine aminotransferase (ALT > 30 U/L, normal <24 U/L).

Exclusion Criteria:

* General exclusion criteria were the presence of other liver disease
* Child B or C cirrhosis
* Severe cardiac or neurological disease
* Co-infection with hepatitis B or HIV
* Hepatocellular carcinoma evaluated by ultrasound and alpha-fetoprotein
* Autoimmune disorders
* Neutrophil count below 1500 per cubic millimetre
* Platelet count below 75000 per cubic millimetre

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HCV-infected Controls, Psychiatric patients, Patients with former drug addiction and patients with methadone substitution
Enrollment: 81 (Actual)
Dates: Start 1999-08; Primary Completion 2002-02 (Actual); Study Completion 2002-05 (Actual)

PRIMARY OUTCOMES:
Response
Sustained Virological Response
Adherence
Occurrence of depression
Occurrence of other psychiatric side effects
Long term outcome

SECONDARY OUTCOMES:
Psychiatric side effects (group comparison)
Long term outcome after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Martin Schaefer, MD, Principal Investigator — Kliniken Essen-Mitte
Locations (1):
- Department of Psychiatry, Munich, Germany

REFERENCES:
- [Result] Schaefer M, Schmidt F, Folwaczny C, Lorenz R, Martin G, Schindlbeck N, Heldwein W, Soyka M, Grunze H, Koenig A, Loeschke K. Adherence and mental side effects during hepatitis C treatment with interferon alfa and ribavirin in psychiatric risk groups. Hepatology. 2003 Feb;37(2):443-51. doi: 10.1053/jhep.2003.50031. PMID 12540795